CLINICAL TRIAL: NCT00732121
Title: Effects of Sitagliptin On Markers of Bone Turnover in Patients With Type 2 Diabetes
Brief Title: Bone Turnover in Type 2 Diabetes Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Richard Pratley, MD, University of Vermont College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Merck-33283
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Sitagliptin
  Interventions: Drug: Sitagliptin
- 2 (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100 mg daily for 4 weeks
  Other Names: Januvia (brand name for sitagliptin)
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Background:

Incretin hormones are hormones produced by the gut in response to food intake. These hormones help the body to control the metabolism of glucose (sugar). In particular, two incretin hormones (GLP-1 and GIP) cause the pancreas to secrete more insulin in response to high blood glucose levels. This helps the body to metabolize the glucose more effectively, lowering blood sugar levels. In addition to their effects on the pancreas, GLP-1 and GIP have effects on other tissues, including the brain, gut, fat cells and bone. A new class of oral drugs developed for the treatment of type 2 diabetes mellitus (T2DM) called DPP-4 inhibitors increases levels of the active forms of GLP-1 and GIP in the body by preventing their breakdown. This study tests whether a medicine in this class called sitagliptin (Januvia), which is commonly used to treat T2DM, affects markers of bone turnover in patients with T2DM. The hypothesis is that treatment with sitagliptin will increase markers of bone formation and decrease markers of bone resorption during a mixed meal, by enhancing active circulating levels of GLP-1, GIP and GLP-2.

Methods:

To address this question we will recruit patients with T2DM whose diabetes is controlled with either diet+exercise or with metformin (another medicine commonly used to treat T2DM). Subjects will undergo measurement of body fat and bone mineral density by DEXA scanning and a 3-hour mixed meal test. During the mixed meal test blood samples will be taken to measure how much GLP-1 and GIP are produced. Markers of bone formation will also be measured in blood samples obtained during the mixed meal test. Subjects will then be randomly assigned to 8 weeks of treatment with either sitagliptin (100 mg/day) or matching placebo (an inactive tablet that does not contain medication). Subjects will be seen 4 weeks after commencing treatment to assess safety and tolerability. After 8 weeks of treatment the meal test will be repeated. Subjects will then be washed off of their initial treatment (sitagliptin or placebo) for 1 week (that is, they will receive no study medication during this period). After the washout period, they will commence a second 8-week period of treatment with the other study medication (that is, if they received sitagliptin initially, they will receive placebo during period 2 and vice-versa). At the end of period 2, subjects will undergo a third mixed meal test with measurement of GLP-1, GIP and markers of bone turnover.

Significance:

Recent studies suggest that oral antidiabetic medications of the thiazolidinedione class, such as rosiglitazone (Avandia) and pioglitazone (Actos), may weaken bones, increasing the risk of fractures in older women with diabetes. The proposed study will test whether drugs of the DPP-4 inhibitor class, such as sitagliptin (Januvia), have beneficial effects on bone turnover by increasing the activity of GLP-1 and GIP. Results of this pilot study may suggest the need to perform longer-term studies to determine whether DPP-4 inhibitors increase bone mineral density and reduce the risk of fractures in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with diet/exercise or metformin
* HbA1c less than or equal to 7%
* Men and women aged 45-80 years old
* If female, must be post-menopausal (natural or surgical)

Exclusion Criteria:

* Endocrine disorders (acromegaly, anorexia, Cushings, type 2 diabetes, hyperparathyroidism, hyperthyroidism, hypercalcemia)
* GI conditions (celiac sprue, gastric bypass/gastrectomy, active inflammatory bowel disease, cirrhosis)
* Cancer (including multiple myeloma) within 3 years of the study (except local non-melanoma skin cancers and cervical carcinoma in situ)
* Active alcoholism or drug abuse
* Chronic kidney disease with a GFR < 60
* HIV/AIDS
* History of hypersensitivity reaction to sitagliptin or other DPP-4 inhibitors
* Hemoglobin < 12 mg/dL for men and < 10 for women
* Taking medications that could affect bone turnover (estrogen, progesterone, testosterone, bisphosphonates, SERMS, calcitonin, teriparatide cyclosporine glucocorticoids, methotrexate or phenothiazines), thiazolidinediones, sulfonylureas, dipeptidyl peptidase-4 inhibitors, exenatide, insulin, weight loss drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-06 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the integrated response to the mixed meal test of markers of bone turnover following 8 weeks of treatment with sitagliptin vs. placebo. | 8 weeks per subject

SECONDARY OUTCOMES:
Change in the active GIP in response to the mixed meal test | 8 weeks
Change in the active GLP-1 in response to the mixed meal test. | 8 weeks
Change in the active GLP-2 in response to the mixed meal test. | 8 weeks
Change in glucose response during the mixed meal test. | 8 weeks
Change in insulin secretion during the mixed meal test. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Pratley, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, South Burlington, Vermont, United States